CLINICAL TRIAL: NCT03484416
Title: Routine Low-dose Calcium and Vitamin D Supplementation for Preventing Symptomatic Postthyroidectomy Hypocalcemia
Brief Title: Routine Calcium for Preventing Hypocalcemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Hyungju Kwon, Assistant Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Rouine Calcium
Record Dates: First submitted 2018-03-25; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Thyroid Neoplasm
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Calcium Carbonate; Vitamin D

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine calcium (Active Comparator): Patients in the routine calcium group received oral supplements of 1,500 mg/day elemental calcium (by calcium carbonate) and 1,000 IU/day cholecalciferol for 2 weeks, beginning on the first postoperative day
  Interventions: Drug: Calcium Carbonate 1500 Mg with Vitamin D
- control (No Intervention): Patients in the control group did not receive calcium or cholecalciferol for 2 weeks

INTERVENTIONS:
Drug: Calcium Carbonate 1500 Mg with Vitamin D — Patients in the routine calcium group received oral supplements of 1,500 mg/day elemental calcium and 1,000 IU/day cholecalciferol (Dicamax 1000) for 2 weeks, whereas control group did not
  Other Names: Dicamax 1000
  Arms: Routine calcium

SUMMARY:
The present study investigated the effect of routine calcium and vitamin D supplementation and tried to find the predictors for postoperative hypocalcemia in patients with thyroid cancer.

DETAILED DESCRIPTION:
The present study investigated the effect of routine calcium and vitamin D supplementation and tried to find the predictors for postoperative hypocalcemia in patients with thyroid cancer. Demographic data, including age, sex, pathologic features, and postoperative laboratory test results were analyzed, as was the development of symptomatic hypocalcemia, defined as an ionized calcium concentration below 4.6 mg/dL (normal range, 4.6-5.4 mg/dL) associated with hypocalcemic symptoms. Hypocalcemia was considered permanent in patients who required calcium supplementation for longer than 6 months after thyroidectomy.

Serum concentrations of PTH and ionized calcium were measured 1 and 14 days postoperatively. Patients in the routine calcium group received oral supplements of 1,500 mg/day elemental calcium and 1,000 IU/day cholecalciferol for 2 weeks, beginning on the first postoperative day (POD) to the 14th POD, whereas patients in the control group received no supplementation. If symptomatic hypocalcemia developed, patients in both groups received 2.0 g of intravenous calcium, followed by oral supplementation with 3,000-4,000 mg/day elemental calcium and 1,000-2,000 IU/day cholecalciferol up to the 14th POD. If hypocalcemic symptoms were persistent or worsening 2 hours after calcium administration, patients were administered another intravenous calcium supplementation.

ELIGIBILITY:
Inclusion Criteria:

* patients with thyroid cancer
* euthyroid state
* underwent total thyroidectomy

Exclusion Criteria:

* previous history of neck surgery or irradiation
* calcium supplement before enrollment
* hyperthyroidism or hypothyroidism
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
symptomatic hypocalcemia | postoperative day 1
  Symptomatic hypocalcemia was defined as an ionized calcium concentration below 4.6 mg/dL (normal range, 4.6-5.4 mg/dL) associated with hypocalcemic symptoms.
permanent hypocalcemia | postoperative 6 months
  Symptomatic hypocalcemia was defined as an ionized calcium concentration below 4.6 mg/dL (normal range, 4.6-5.4 mg/dL) associated with hypocalcemic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Hyungju Kwon, MD, Principal Investigator — Ewah Womans University Medical Center
Locations (1):
- Ewha Womans University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No